CLINICAL TRIAL: NCT06290284
Title: Comparison Between the Long (Mini-midline) and the Short Catheter (Peripheral Intravenous Catheter) in the Reduction of Venipunctures During Hospital Stay: a Randomized Controlled Trial
Brief Title: Comparison Between Mini-midline and the Peripheral Intravenous Catheter
Acronym: INSERT/2022
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Alessandro Galazzi, Principal investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6322
Record Dates: First submitted 2024-01-31; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Vascular Access Devices; Venous Puncture
Keywords: Vascular access; Emergency Department; Long Peripheral Catheter; Peripheral Intra-Venous Catheter
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician will be provided an anonymized dataset.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long Peripheral Catheter (Experimental): The procedure to place a LPC includes these steps: before inserting the catheter, the nurse will perform routine preliminary (non sterile) inspection of the arm to identify an insertion site. After selecting the insertion site, the nurse will release the tourniquet, with non-sterile gloves, and disinfect the skin around the insertion site. While allowing the antiseptic to act, the nurse will apply the tourniquet, and pull lightly with the thumb of the non-dominant hand to keep the vein from moving. After the needle has been inserted in the vein lumen, the guide wire is advanced and the catheter is inserted using the catheter wings. As the catheter is being inserted, the sheath (housing) is removed and then the wings. Before attaching the catheter to an extension without a needle or to a 3-way stopcock, it should be connected to a statlock to ensure it is safely fixated. A transparent, semi-permeable dressing will allow for daily visual inspection of the insertion site.
  Interventions: Procedure: Long Peripheral Catheter
- Peripheral Intra-Venous Catheter (Active Comparator): The procedure to place a PIVC includes these steps: before inserting the catheter, the nurse will perform routine preliminary (non sterile) inspection of the arm to identify an insertion site. After selecting the insertion site, the nurse will release the tourniquet, with non-sterile gloves, and disinfect the skin around the insertion site. While allowing the antiseptic to act, the nurse will apply the tourniquet, and pull lightly with the thumb of the non-dominant hand to keep the vein from moving. The needle will be inserted at a 10-30 degree angle about 1-2 cm distal from the catheter insertion site. Holding the needle firmly, the nurse will advance the cannula for its entire length into the lumen, remove the needle, and connect the cannula via an extension to a 3-way stopcock. A transparent, semi-permeable dressing will allow for daily visual inspection of the insertion site.
  Interventions: Procedure: Peripheral Intra-Venous Catheter

INTERVENTIONS:
Procedure: Long Peripheral Catheter — PowerGlide Pro™ Midline Catheter
  Arms: Long Peripheral Catheter
Procedure: Peripheral Intra-Venous Catheter — Venflon™ Pro Safety Needle Protected IntraVenous Cannula
  Arms: Peripheral Intra-Venous Catheter

SUMMARY:
The goal of this randomized controlled trial is to investigate the difference between LPC (mini-midline) and PIVC (peripheral venous catheter) on the need of further venipuncture for blood withdrawal or placement of a new vascular access.

The main questions it aims to answer are:

* Whether the number of patients with LPC and PIVC differ in terms of repeated venipunctures;
* Whether the number of patients with LPC and PIVC differ in terms of adverse events associated with the use of such vascular catheters.

Researchers will compare the proportion of patients with repeated venipunctures between LPC and PIVC arms.

DETAILED DESCRIPTION:
A standard peripheral intravenous catheter (PIVC) or a mini-midline (LPC) will be placed according to routine clinical indications (i.e., for blood withdrawal and IV drug therapy) in patients seeking care at the Emergency Department. On admission at the Emergency Department triage desk, patients will be assigned a triage code according to clinical assessment by the triage nurse and will be evaluated as to the probability of being eventually admitted to hospital. Following enrollment, patients will be randomly assigned to receive LPC or PIVC. The follow-up period begins after catheter placement and continues through transfer to a hospital ward. During this period of catheter management, the insertion site and dressing will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* High probability of hospital admission
* Sufficient venous patrimony according to EA-DIVA scale score

Exclusion Criteria:

* Patients already having a venous access in place
* Patients requiring life-saving treatments
* Patients seeking ambulatory care
* Patients unable to express informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Difference in proportion | The catheter will be evaluated within 24 hours after the placement
  Difference between the two study arms in the proportion of patients who required a venipuncture after insertion of the PIVC or the LPC.

SECONDARY OUTCOMES:
Adverse events associated with use of LPC and PIVC | Adverse will be evaluated every 24 hours till the catheter removal
  Number of adverse events (e.g., thrombophlebitis, extravasation, inflammation of the insertion site) monitored also using the Visual Infusion Phlebitis Score

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Galazzi, PhD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Civetta G, Cortesi S, Mancardi M, De Pirro A, Vischio M, Mazzocchi M, Scudeller L, Bottazzi A, Iotti GA, Palo A. EA-DIVA score (Enhanced Adult DIVA score): A new scale to predict difficult preoperative venous cannulation in adult surgical patients. J Vasc Access. 2019 May;20(3):281-289. doi: 10.1177/1129729818804994. Epub 2018 Oct 16. PMID 30324841
- [Derived] Binda F, Galazzi A, Marelli F, Salinaro G, de Vecchi M, Spagna S, Marcotullio A, Calegari J, Laquintana D, Gambazza S. Long versus conventional peripheral intravenous catheters to reduce venipunctures during hospital stay: A randomized controlled trial. J Vasc Access. 2025 Nov 3:11297298251385595. doi: 10.1177/11297298251385595. Online ahead of print. PMID 41185485